CLINICAL TRIAL: NCT05165732
Title: A Randomized, Open, Control Phase ⅠV Clinical Trial, to Evaluate One Booster Immunization of Inactivated COVID-19 Vaccine (CoronaVac) or Original Vaccine in Adults Aged 18-45 Years Old Previously Vaccinated With Inactivated COVID-19 Vaccine From Difference Manufactures
Brief Title: Safety and Immunogenicity Study of Booster Vaccination With COVID-19 Vaccine (Vero Cell),Inactivated From Different Manufactures for Prevention of COVID-19
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Limited subjects
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-nCOV-4012
Record Dates: First submitted 2021-12-20; First posted 2021-12-21 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Experimental Group 1 (Experimental): 96 subjects who completed primary immunization with inactivated COVID-19 vaccine manufactured by Sinovac Research & Development Co.,Ltd. will receive one dose of booster immunization with inactivated COVID-19 vaccine manufactured by Sinovac Research & Development Co.,Ltd.
  Interventions: Biological: Experimental vaccine 1
- Experimental Group 2 (Experimental): 96 subjects who completed primary immunization with inactivated COVID-19 vaccine manufactured by Beijing institute of Biological Products Co,Ltd. will receive one dose of booster immunization with inactivated COVID-19 vaccine manufactured by Sinovac Research & Development Co.,Ltd.
  Interventions: Biological: Experimental vaccine 1
- Experimental Group 3 (Experimental): 96 subjects who completed primary immunization with inactivated COVID-19 vaccine manufactured by Beijing institute of Biological Products Co.,Ltd. will receive one dose of booster immunization with inactivated COVID-19 vaccine manufactured by Beijing institute of Biological Products Co.,Ltd.
  Interventions: Biological: Experimental vaccine 2
- Experimental Group 4 (Experimental): 92 subjects who completed primary immunization with inactivated COVID-19 vaccine manufactured by Wuhan Institute of Biological Products Co.,Ltd will receive one dose of booster immunization with inactivated COVID-19 vaccine manufactured by Sinovac Research & Development Co.,Ltd.
  Interventions: Biological: Experimental vaccine 1
- Experimental Group 5 (Experimental): 92 subjects who completed primary immunization with inactivated COVID-19 vaccine manufactured by Wuhan Institute of Biological Products Co.,Ltd will receive one dose of booster immunization with inactivated COVID-19 vaccine manufactured by Wuhan Institute of Biological Products Co.,Ltd.
  Interventions: Biological: Experimental vaccine 3

INTERVENTIONS:
Biological: Experimental vaccine 1 — Inactivated COVID-19 vaccine manufactured by Sinovac Life Sciences Co., Ltd.600SU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection.
  Arms: Experimental Group 1; Experimental Group 2; Experimental Group 4
Biological: Experimental vaccine 2 — Inactivated COVID-19 vaccine manufactured by Beijing Institute of Biological Products Co.,Ltd.4ug inactivated virus in 0.5 mL of aluminium hydroxide solution per injection.
  Arms: Experimental Group 3
Biological: Experimental vaccine 3 — Inactivated COVID-19 vaccine manufactured by Wuhan Institute of Biological Products Co.,Ltd.200WU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection.
  Arms: Experimental Group 5

SUMMARY:
This is a randomized, Open, control phase Ⅳ clinical trial of inactivated COVID-19 vaccine manufactured by Sinovac Research & Development Co., Ltd,Beijing institute of Biological Products Co.,Ltd and Wuhan Institute of Biological Products Co.,Ltd.The purpose of this study is to explore booster Immunization of SARS-CoV-2 Inactivated Vaccine from different manufactures in adults aged 18-45 years old Previously Vaccinated with inactivated COVID-19 vaccine

DETAILED DESCRIPTION:
This study a randomized, Open, control phase Ⅳclinical trial of inactivated COVID-19 vaccine .The purpose of this study is to explore booster Immunization of SARS-CoV-2 inactivated vaccine from different manufactures in adults aged 18-45 years old previously vaccinated with inactivated COVID-19 vaccine.A total of 480 subjects who have completed vaccination of two doses of inactivated COVID-19 vaccine for 6 to 8 months will be enrolled.In this study ,96 subjects who completed primary immunization with inactivated COVID-19 vaccine manufactured by Sinovac Research & Development Co.,Ltd. will receive one dose of booster immunization with inactivated COVID-19 vaccine manufactured by Sinovac Research & Development Co.,Ltd.(experimental group 1).192 subjects who completed primary immunization with inactivated COVID-19 vaccine manufactured by Beijing institute of Biological Products Co.,Ltd. will be randomly divided into two groups (experimental group 2 and experimental group 3) in a 1:1 ratio and receive one dose of booster immunization with inactivated COVID-19 vaccine manufactured by Sinovac Research & Development Co.,Ltd. and Beijing institute of Biological Products Co., Ltd,respectively.192 subjects who completed primary immunization with inactivated COVID-19 vaccine manufactured by Wuhan Institute of Biological Products Co.,Ltd.will be randomly divided into two groups(experimental group 4 and experimental group 5) in a 1:1 ratio and receive one dose of booster immunization with inactivated COVID-19 vaccine manufactured by Sinovac Research & Development Co.,Ltd. and Wuhan Institute of Biological Products Co.,Ltd.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-45;
* Proven legal identity;
* The subjects can understand and voluntarily sign the informed consent form and be willing to complete the study in accordance with the study plan;
* Have completed two doses of SARS-CoV-2 inactivated vaccine vaccination for 6 to 8 months(the interval between the two doses vaccine of primary immunization is 21~35 days, and the two doses vaccine of primary immunization should be manufactured by the same manufactures).

Exclusion Criteria:

* History of SARS-CoV-2 infection(laboratory confirmed);
* Have received inactivated SARS-CoV-2 vaccine from other manufacturers other than Sinovac Life Sciences Co., Ltd.,Beijing Institute of Biological Products Co.,Ltd.and Wuhan Institute of Biological Products Co.,Ltd.and received three and more doses of inactivated SARS-CoV-2 vaccine;
* Severe adverse reactions, such as urticaria, dyspnea, and angioneurotic edema , occurred during the primary immunization;
* Autoimmune disease such as systemic lupus erythematosus or immunodeficiency / immunosuppression such as AIDS, post-transplant;
* Severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver or kidney diseases, malignant tumors, etc;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids(excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* History of alcohol or drug abuse;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Acute diseases or acute exacerbation of chronic diseases within 7 days prior to booster vaccination;
* Axillary temperature >37.0°C;
* Already pregnant or are breastfeeding, planning to get pregnant within

  1months (according to subjects' self-report and urine pregnancy test results);
* Participated in other clinical trials prior to enrollment and during the followup period, or planned to participate in other clinical trials during the clinical trial period;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2023-03-20 (Estimated); Study Completion 2023-08-20 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity index-GMT of neutralizing antibodies | 28 days after booster dose
  GMT of neutralizing antibody 28 days after booster dose.
Immunogenicity index-seroconversion rate (4-fold and above increase)of neutralizing antibodies | 28 days after booster dose
  Seroconversion rate (4-fold and above increase)of neutralizing antibodies 28 days after booster dose.
Immunogenicity index-seropositive rate of neutralizing antibody | 28 days after booster dose
  Seropositive rate of neutralizing antibody 28 days after booster dose.

SECONDARY OUTCOMES:
Safety index-Incidence of adverse reactions | 0-28 days after booster
  Incidence of adverse reactions occured 0-28 days after booster
Safety index-Incidence of adverse reactions | 0-7 days after booster dose
  Incidence of adverse reactions occurred 0-7 days after booster dose.
Safety index-Incidence of SAEs and AESIs | 0-28 days after booster
  Incidence of SAEs and AESIs occured 0-28 days after booster.

CONTACTS AND LOCATIONS:
Overall Officials: Qiuyue Mu, Master, Principal Investigator — Guizhou Provincial Center for Disease Prevention and Control
Locations (1):
- Yanhe Tujia Autonomous County Center for Disease Control and Prevention, Tongren, Guizhou, China